CLINICAL TRIAL: NCT02517229
Title: The Effect of Altered Gravity Condition on Postural Control
Acronym: POSTURGRAV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-084
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- in balance control in response to microgravity (Other): to evaluate changes in balance control in response to microgravity during reactive balance tasks compared to normal gravity.
  Interventions: Other: Parabolic flight; Other: balance control measurements; Device: electromagnetic maneuverable postural platform

INTERVENTIONS:
Other: Parabolic flight
Other: balance control measurements
Device: electromagnetic maneuverable postural platform

SUMMARY:
The scientific goal of this experiment is to evaluate changes in balance control in response to microgravity during reactive balance tasks. For that purpose, kinematic and neuromuscular parameters under microgravity are compared to normal gravity conditions. To induce postural responses among the test subjects, an electromagnetic maneuverable postural platform will be used in order to randomly elicit perturbations. Postural reactions will be quantified by means of mechanical and electromyographic data. In Addition, peripheral nerve stimulation will be used to assess the spinal excitability by means of H-reflex recordings. H-reflex measurements were chosen as they allow reliable information about inhibitory and facilitatory mechanisms taking place at the spinal level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 21 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with medical history of neurological disorders
* Person with medical history of musculoskeletal disorders of the lower limbs, especially of the ankle and knee joint.
* Pregnant women

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
balance skill, expressed by the postural sway in mm | baseline
neuromuscular activity, expressed by the Electromyograpy (EMG)-amplitudes | baseline
spinal excitability, expressed by H-Reflexes | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France